CLINICAL TRIAL: NCT04504084
Title: Influence of Patient Decision-Making Aids for Patients With Unilateral Ureteral Stone: A Randomized-Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N202003100
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Patient Decision Aids; Ureteral Stone; Shared Decision Making
MeSH Terms: conditions — Ureterolithiasis | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid group (Experimental): Shared decision making using decision aid
  Interventions: Other: Decision aid
- Controlled group (No Intervention): Standard oral explanation the details of treament options

INTERVENTIONS:
Other: Decision aid — Patient Decision Aid is a tool that helps patient with ureteral stone become involved in decision making on choosing treatment for ureteral stone. Patient Decision Aid provides information about the options and outcomes, and by clarifying personal values.
  Arms: Decision aid group

SUMMARY:
Ureteral stone is a common disease with high prevalence and recurrence rate in Taiwan. Taiwan is located in subtropical zone, where urolithiasis is commonly seen. A national survey in Taiwan determined that 9.6% of the population suffered stones throughout their lifetime. Symptoms of ureteral stone include renal colic, hematuria, and urinary tract infection. Without proper treatment, ureteral stone could lead to renal function impairment such as acute kidney injury (AKI) or chronic kidney disease (CKD). There are several treatment options for ureteral stone, such as ureteroscopic lithotripsy (URSL), flexible urteroscopic lithotripsy (F-URSL), percutaneous nephrolithotomy (PCNL), extracorporeal shock wave lithotripsy (ESWL), and Medical expulsive therapy (MET).

However, there are only few minutes from diagnosis of ureteral stone to possible treatment options explanation. It's difficult for patients to well understand all the details of possible treatments under such circumstances.

Therefore, we design a patient decision aid (PDA) for unilateral ureteral stone to help patients understand all the treatment options. The PDA is standardized, written in plain language and patient-centered, with pictures attached.

DETAILED DESCRIPTION:
Background:

Shared decision making (SDM) has been defined as: 'an approach where clinicians and patients share the best available evidence when faced with the task of making decisions, and where patients are supported to consider options, to achieve informed preferences". To conduct SDM, a PDA was developed to be administered for patients with ureteral stone to choose treatment options. We expect the PDA would benefit the intervention group in the aspects of knowledge and communication in choosing treatment.The aim of this study is to conduct a single center randomized controlled trial (RCT ) to evaluate the benefit of PDAs on decision making.

Patients and Methods:

Decision aids are interventions designed to help patients with ureteral stone to choose their treatment options for unilateral ureteral stone and any potential outcome relevant to treatment options. Patients with unilateral ureteral stone are randomly assigned to receive a PDA (PDA group) or the standard oral information (control group) during consultation.

In control group, patients will receive standard oral information. In PDA group group, PDA will be used as a tool to explain the benefits and harms between ureteroscopic lithotripsy (URSL), flexible urteroscopic lithotripsy (F-URSL), extracorporeal shock wave lithotripsy (ESWL). And by following SDM principles, the patients are guided to consider their individual values and preferences and helped to make a choice that best meet their needs. This study will be conducted in a single center (Shuang Ho Hospital). The outcomes are decision conflicts and decision-making and SURE test before treatment.

Hypothesis:

We expect that the PDA would promote communications between doctors and patients, to further help the patient to make a proper decision for his/her own.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 75
* Ureteral stone diagnosed with KUB, IVP or CT
* Stone size between 0 to 2 cm

Exclusion Criteria:

* Stone passage spontaneously
* Patients who do not speak Mandarian
* Patients with dementia
* Nationality not Republic of China
* Patients with bilateral ureteral stone
* Patients with staghorn stone
* Patients with bladder stone
* Patients with severe infection
* Pregnant women
* Others patients could not communicate with

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision conflicts | For patients choose URSL or F-URSL, one day before the operation. For patients choose ESWL, half an hour before the treatment.
  Total score of decisional conflict scale

SECONDARY OUTCOMES:
SURE test | For patients choose URSL or F-URSL, one day before the operation. For patients choose ESWL, half an hour before the treatment.
  Total score of SURE test

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Te Chiang, MD, Principal Investigator — No.291, Zhongzheng Rd., Zhonghe , Taipei 23561, Taiwan. Shuanghe Hospital